CLINICAL TRIAL: NCT04604691
Title: Blinatumomab for Minimal Residual Disease Before Hematopoietic Stem Cell Transplantation With Pediatric B-cell Precursor Acute Lymphoblastic Leukemia
Brief Title: Blinatumomab in Pediatric B-cell Acute Lymphoblastic Leukemia (ALL) With Minimal Residual Disease (MRD)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20197007
Record Dates: First submitted 2020-10-21; First posted 2020-10-27 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Pediatric ALL, B Cell; Minimal Residual Disease
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasm, Residual | interventions — blinatumomab; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Blinatumomab Treatment (Experimental)
  Interventions: Drug: Blinatumomab for Injection

INTERVENTIONS:
Drug: Blinatumomab for Injection — Blinatumomab will be administered as a continuous intravenous (CIV) infusion at a constant flow rate over four weeks followed by a two-week infusion free interval.

SUMMARY:
This is a single-arm, open-label, multi-center phase I study using blinatumomab for pediatric B-cell acute lymphoblastic leukemia patients with positive of minimal residual disease. 1 Cycle of blinatumomab treatment followed by hematopoietic stem cell transplantation. Blinatumomab has approved to treat adults and children with B-cell precursor ALL who are in remission but still have MRD. However, data on the effects and safety of blinatumomab in children with B-precursor ALL with MRD positive are insufficient.

ELIGIBILITY:
Inclusion Criteria:

* Immunophenotypic evidence of Cluster of Differentiation 19 (CD19) positive B precursor ALL
* Age <18 years at the time of informed consent/assent
* B cell precursor ALL in first or later hematologic complete remission (CR) defined as less than 5% blasts in bone marrow after at least three intense chemotherapy blocks
* Persistent or recurrent MRD ≥10^-4 in an assay with a minimum sensitivity of 10^-5 before hematopoietic stem cell transplantation
* Bone marrow function as defined below: Absolute neutrophil count ≥1,000/μL, Platelets ≥50,000/μL (transfusion permitted), Hemoglobin level ≥9 g/dL (transfusion permitted)
* Renal and hepatic function as defined below: Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), and alkaline phosphatase (AP) < 2 x upper limit of normal (ULN), Total bilirubin <1.5 x ULN, Creatinine clearance ≥ 50 mL/min
* Negative HIV test, negative hepatitis B (HBsAg) and hepatitis C virus (anti-HCV) test
* Negative pregnancy test in women of childbearing potential

Exclusion Criteria:

* Presence of circulating blasts or current extramedullary involvement by ALL
* History of relevant central nervous system (CNS) pathology or current relevant CNS pathology (e.g. seizure, epilepsy, paresis, aphasia, stroke, severe brain injuries, dementia, cerebellar disease, organic brain syndrome, psychosis) with the except of CNS leukemia that is well controlled with intrathecal therapy
* Current infiltration of cerebrospinal fluid by ALL
* History of or active relevant autoimmune disease
* Systemic cancer chemotherapy within 2 weeks prior to study treatment (except for intrathecal prophylaxis)
* Radiotherapy within 4 weeks prior to study treatment
* Autologous hematopoietic stem cell transplantation (HSCT) within six weeks prior to study treatment
* Therapy with monoclonal antibodies (rituximab, alemtuzumab) within 4 weeks prior to study treatment
* Treatment with any investigational product within 4 weeks prior to study treatment
* Known hypersensitivity to immunoglobulin or to any other component of the study drug formulation
* Active malignancy other than ALL with the exception of basal cell or squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix
* Active infection, any other concurrent disease or medical condition that are deemed to interfere with the conduct of the study as judged by the investigator

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation including cytokine release syndrome | At the latest possible timepoint prior to the initiation of transplant conditioning or after 30 days of Blinatumomab treatment
  The incidence of treatment-emergent and treatment-related adverse events

SECONDARY OUTCOMES:
Complete MRD response status after 1 cycle of blinatumomab | 28 Days
Hematologic Relapse-Free Survival (RFS) | 24 Months
Overall Survival (OS) | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung Jin Kang, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea